CLINICAL TRIAL: NCT01231685
Title: A Randomized Prospective Open Label Study of Switching to Raltegravir Based ART Compared to Maintaining Ritonavir Boosted PI-based ART on Liver Fibrosis Progression in HIV-HCV Coinfected Patients
Brief Title: Raltegravir Switch Study to Reduce Liver Fibrosis Progression in HIV-Hepatitis C Co-infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); CIHR Canadian HIV Trials Network (Network)
Responsible Party: Principal Investigator, Marina Klein, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTN260
Record Dates: First submitted 2010-10-29; First posted 2010-11-01 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: HIV; Hepatitis C; Liver Fibrosis
Keywords: Liver fibrosis; HIV; Hepatitis C Virus; Coinfection
MeSH Terms: conditions — Hepatitis C; Liver Cirrhosis; Coinfection | interventions — Raltegravir Potassium; lopinavir-ritonavir drug combination; Lopinavir; atazanavir, ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ritonavir-boosted protease inhibitor (Active Comparator)
  Interventions: Drug: Raltegravir; Drug: Ritonavir-boosted protease inhibitor
- Raltegravir (Experimental)
  Interventions: Drug: Raltegravir; Drug: Ritonavir-boosted protease inhibitor

INTERVENTIONS:
Drug: Raltegravir — Subjects will maintain their nucleoside backbone and switch ritonavir-boosted protease inhibitor to Raltegravir 400 mg po BID for 48 weeks.
  Other Names: Isentress; MK-0518; RGV
Drug: Ritonavir-boosted protease inhibitor — Subjects will maintain their nucleoside backbone and remain on a ritonavir-boosted protease inhibitor at standard doses for for 48 weeks
  Other Names: Kaletra; Lopinavir-ritonavir; Atazanavir-ritonavir; Reyataz-norvir; Darunavir-ritonavir; Presista-norvir

SUMMARY:
HIV infection exerts a negative impact on the course of HCV infection. Co-infected individuals progress more rapidly to liver fibrosis, cirrhosis and ESLD compared to those infected with HCV alone. Some of the this accelerated fibrosis may be related to longterm chronic toxicity from protease inhibitor based ART.

Hypothesis: Switching from ritonavir boosted-PI based ART regimen to a Raltegravir-based regimen will reduce the rate of hepatic fibrosis progression in HIV-HCV co-infected patients as measured by transient elastography (Fibroscan®) and the AST-to-platelet ratio index (APRI).

DETAILED DESCRIPTION:
Primary Objective-To assess if switching from ritonavir boosted-PI based ART regimen to a Raltegravir-based regimen will reduce the rate of hepatic fibrosis progression in HIV-HCV co-infected patients as measured by transient elastography (Fibroscan®) and the AST-to-platelet ratio index (APRI) after 48 weeks of treatment.

Secondary Objectives:

(i) To assess the safety and tolerability of switching from a ritonavir boosted-PI ART regimen to a raltegravir-based regimen for 48 weeks.

(ii) To evaluate hepatic function (liver enzymes) at weeks 0, 2, 4, 8, 12, 24, 36, 48 and 72 post switch.

(iii) To evaluate the effect of switching treatment on control of HIV infection (as measured by HIV viral load and CD4) at weeks 0, 4, 8, 12, 24, 36, 48, and 72 post switch.

(iv) To evaluate metabolic profiles (e.g, fasting lipid profiles, glucose and insulin) at weeks 0, 24, 48 and 72 post switch.

(v) To evaluate inflammatory markers associated with liver fibrosis at weeks 0, 2, 4, 8, 12, 24, 36, 48 and 72 post switch.

Population: Patients will be selected from CTN222; a Canadian National multisite prospective cohort of HCV-HIV infected persons (N=978) or from other eligible patients followed at participating sites. All patients recruited into the cohort are adults aged over 16 years old with documented HIV infection (ELISA with western blot confirmation) and with chronic HCV infection or evidence of HCV exposure (e.g. HCV-seropositive by ELISA with RIBA II or EIA confirmation, or if serologically false negative, HCV RNA+).

Study Design: A Randomized Prospective Open label study

Sample Size:

N = 40 This is a Phase II study designed to evaluate the safety and feasibility of a switch to raltegravir in HIV-HCV co-infected patients. As neither the duration of time required to improve fibrosis nor the potential impact of such a switch currently is known, this trial will provide important pilot data with which to estimate the true effect size and calculate the sample size required to conduct a larger definitive study on this question. It is hypothesized that switching therapy will lead to significant reduction in fibrosis as measured by APRI and FibroScan®. In other studies, for example, of successful HCV treatment using FibroScan®, a 34% reduction in fibrosis score was observed in those obtaining a sustained virologic response at 48 weeks (e.g., from mean baseline score of 10.3 kPa to 6.6 kPa at 48 weeks; s.d.= 5 kPa 1). We propose a sample size of 20 patients in each group, which would provide approximately 80% power to detect at least a difference of 5 kPa in fibrosis score change between the two groups assuming a similar standard deviation.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older
2. Chronic HIV-HCV co-infection (HCV RNA + for at least 6 months and could have had previous HCV treatment).
3. Receiving ritonavir boosted PI-based ART for at least 6 months.
4. APRI score ≥ 1.5 (equivalent to liver biopsy score of ≥ F2) AND/OR Fibroscan > 6.9KPa
5. HIV viral suppression (<50 copies/mL) for at least 6 months.
6. No prior evidence of resistance to raltegravir or co-administered nucleoside backbone.
7. No prior history of virologic failure.

Exclusion Criteria:

1. Clinical evidence of decompensated liver disease (e.g., ascites, esophageal varices, or hepatic encephalopathy hepatoma or hepatocellular carcinoma).
2. Chronic Hepatitis B infection (defined as positive HBsAg or Hepatitis B viral load greater than 10,000 copies/mL).
3. AFP greater than or equal to 200 ng/mL at screening.
4. Known or suspected Wilson's disease, alpha-1-antitrypsin deficiency, celiac disease or other cause of chronic liver disease.
5. Chronic renal insufficiency (eGFR < 20 mL/min) at screening.
6. Pregnancy and planned pregnancy (WOCBP not using adequate contraception).
7. Women who are breastfeeding.
8. Active opportunistic infection (except oral thrush) or neoplasm (except Kaposi's sarcoma, skin cancer, or cancer of the cervix or anus, unless known or suspected liver metastasis).
9. Patients intending to start HCV therapy within the treatment phase (within the year following the baseline visit).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2011-12; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of switch on change in liver fibrosis score | 48 weeks
  Change in fibrosis will be assessed by:
  1. Change in Fibroscan® score (kPa) at 48 weeks from baseline
  2. Change in log transformed AST-to-platelt ratio (APRI) score at 48 weeks from baseline

SECONDARY OUTCOMES:
To evaluate inflammatory markers associated with liver fibrosis | 72 weeks
  As a switch from protease inhibitors based regimen to a raltegravir based regimen may impact the liver through various potential mechanisms, we will explore the impact of treatment switching on inflammatory biomarkers.
To evaluate effect of switch on hepatic function | 72 weeks
  Liver enzymes, albumin, direct bilirubin and INR will be measured at week 0,2,4,8,12,24,36,40 and 72.
To evaluate effect of switch on metabolic parameters | 72 weeks
  Metabolic parameters, such as fasting glucose, lipid and insulin profiles will be measured at week 0,24 and 48 post switch
Immunologic and virologic safety | 72 weeks
  To ensure safety, with respect to control of HIV infection following a switch to raltegravir, HIV viral load and CD4 cell counts will be measured at weeks 0,4,8 12, 24, 36, 48 and 72 post switch.

CONTACTS AND LOCATIONS:
Overall Officials: Marina B Klein, MD. M.Sc., Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (3):
- Canada (3):
  - Providence Health Care- St. Paul's Hospital, Vancouver, British Columbia
  - University Health Network - Toronto General Hospital Division, Toronto, Ontario
  - Montreal Chest Institute, Montreal, Quebec

REFERENCES:
- [Background] Vispo E, Mena A, Maida I, Blanco F, Cordoba M, Labarga P, Rodriguez-Novoa S, Alvarez E, Jimenez-Nacher I, Soriano V. Hepatic safety profile of raltegravir in HIV-infected patients with chronic hepatitis C. J Antimicrob Chemother. 2010 Mar;65(3):543-7. doi: 10.1093/jac/dkp446. Epub 2009 Dec 23. PMID 20032006
- [Background] Eron JJ, Young B, Cooper DA, Youle M, Dejesus E, Andrade-Villanueva J, Workman C, Zajdenverg R, Fatkenheuer G, Berger DS, Kumar PN, Rodgers AJ, Shaughnessy MA, Walker ML, Barnard RJ, Miller MD, Dinubile MJ, Nguyen BY, Leavitt R, Xu X, Sklar P; SWITCHMRK 1 and 2 investigators. Switch to a raltegravir-based regimen versus continuation of a lopinavir-ritonavir-based regimen in stable HIV-infected patients with suppressed viraemia (SWITCHMRK 1 and 2): two multicentre, double-blind, randomised controlled trials. Lancet. 2010 Jan 30;375(9712):396-407. doi: 10.1016/S0140-6736(09)62041-9. Epub 2010 Jan 12. PMID 20074791